CLINICAL TRIAL: NCT05394324
Title: A Post-market Clinical Study to Collect Safety and Performance Data on Johnson & Johnson Surgical Vision Products
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JJSV301PMCF
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Refractive Error; Glaucoma; Cataracts; Clear Lens Exchange
MeSH Terms: conditions — Refractive Errors; Glaucoma; Cataract | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intervention — No study treatments will be administered during this retrospective study. However, data will be collected from medical records of patients who have been treated with subject devices of this study.

SUMMARY:
Retrospective collection of data from medical records, multicenter, post-market clinical follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been implanted with and/or undergone ophthalmic surgery using targeted JJSV products
2. Status post ophthalmic surgery between 1 day and 24 months for Year 1. Subsequent years after Year 1 will be between 1 day and 18 months.

Exclusion Criteria:

1. Concurrent participation (during the retrospective follow-up period) in an interventional (drug, device, biologic, etc.) clinical trial
2. Use of surgical devices not in accordance with the product labeling or indications for use
3. Degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that cause visual acuity losses to a level worse than 0.2 logMAR (0.63 decimal, 6/9.5 or 20/32 Snellen) during the retrospective data collection period
4. Use of systemic or ocular medications that may affect vision during the retrospective data collection period
5. Known ocular disease or pathology that, in the opinion of the investigator may confound study findings during the retrospective data collection period
6. Pregnancy, lactating, or other condition associated with hormonal fluctuation that could lead to refractive changes during the retrospective data collection period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been implanted with and/or have undergone ophthalmic surgery using commercial JJSV product(s).
Sampling Method: Non-Probability Sample
Enrollment: 1674 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to 12 months post-operation
  incidence of adverse events that are specified in the ISO 11979-7 Safety and Performance Endpoints.
BCDVA | up to 12 months post-operation
  The proportion of eyes achieving 20/40 or better BCDVA.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (13):
- United States (4):
  - Trinity Research Group, LLC, Dothan, Alabama
  - Empire Eye and Laser Center, Bakersfield, California
  - Chu Vision Institute, Bloomington, Minnesota
  - Valley Retina Institute, McAllen, Texas
- Germany (3):
  - Augenaerzte Gerl & Kollegen MVZ Ahaus GmbH, Ahaus, North Rhine-Westphalia
  - Augenzentrum Erzgebirge, Zschopau, Saxony
  - Augentagesklinik Spreebogen Berlin GbR, Berlin
- Spain (6):
  - Clinica Vistahermosa, Alicante, Alacant
  - Hospital La Arruzafa, Córdoba, Andalusia
  - Instituto Universitario de Oftalmobiologia Aplicada, Valladolid, CL
  - Hosp. De La Santa Creu I Sant Pau, Barcelona, CT
  - Hospital Clinico San Carlos, Madrid, MD
  - Clinica Oftalvist, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu